CLINICAL TRIAL: NCT03737721
Title: UNresectable Squamous Cell Carcinoma Treated With Avelumab and Radical Radiotherapy. A Study to Evaluate the Efficacy and Safety of the Combined Use of Avelumab With Radiation Therapy for the Treatment of Unresectable Cutaneous Squamous Cell Carcinoma
Brief Title: The UNSCARRed Study: UNresctable Squamous Cell Carcinoma Treated With Avelumab and Radical Radiotherapy
Acronym: UNSCARRed
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Loss of Pharma Support
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: EMD Serono (Industry); Alberta Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNSCARRed: IIT-0004
Record Dates: First submitted 2018-10-26; First posted 2018-11-09 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Squamous Cell Carcinoma of the Skin
MeSH Terms: interventions — avelumab

STUDY DESIGN:
Intervention Model Description: This study has been designed as an open-label, non-randomized, single-arm phase II study to investigate the feasibility and efficacy of Avelumab in combination with radiation therapy in patients with unresectable cuSCC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Avelumab and Radical radiotherapy (Experimental): Single-arm combining Avelumab with radical radiotherapy.
  Interventions: Combination Product: Avelumab and Radical radiotherapy

INTERVENTIONS:
Combination Product: Avelumab and Radical radiotherapy — A single-arm, interventional study combining Avelumab with radical radiotherapy. Avelumab will be delivered on a 14-day cycle, with the first cycle administered 14 days in advance of the radiation therapy start date; 63-66 Gy radiation will be delivered over 30 daily fractions concurrent with an additional 4 cycles of Avelumab

SUMMARY:
The purpose of this study is to find out what effects the combination of radiation therapy and Avelumab have on you and your cancer. The effectiveness of this treatment as well as what side effects occur will both be studied.

Squamous cell carcinoma of the skin is the most commonly diagnosed cancer. Risk factors for the development of squamous cell cancer include ultraviolet (sun) exposure, as well as increasing age. In the majority of instances, a minor surgical procedure is curative. Less commonly, squamous cell carcinoma cannot be removed surgically, due to the location and/or extent of the cancer, or due to patient-specific factors which would make surgery unsafe (for instance, the presence of unrelated medical illnesses such as heart disease or stroke).

When squamous cell carcinoma cannot be removed surgically, radiation therapy may serve as an effective alternative treatment. Squamous cell carcinomas are typically very sensitive to radiation, and in some instances radiation therapy may also cure a person of their cancer.

While some people may be cured by radiation therapy, not all people are. This study is investigating the combination of radiation therapy and immune therapy. When given together, more patients may be cured of their cancer.

Immune therapy is effective for the treatment of squamous cell carcinoma. In clinical trials, more than half of patients benefit from immune therapy. Immune therapy is not chemotherapy. Instead, immune therapy involves the infusion of antibodies which target a person's own immune system. Immune therapy "re-activates" a person's own immune system against their cancer.

The treatment offered within this clinical trial includes daily radiation treatments as well as immunotherapy treatments administered once every two weeks. The immunotherapy in use is a drug called Avelumab, which is an antibody that helps your body's immune system fight cancer.

Health Canada, the regulatory body that oversees the use of natural health products, drugs and devices in Canada, has not approved the sale or use of this product to treat this kind of cancer, although they have allowed its use in this study

DETAILED DESCRIPTION:
The treatment of patients with unresectable cuSCC is challenging, and represents an area of high unmet need. Treatment options within this patient population are limited; hence most patients undergo monotherapy with radiation leading to suboptimal outcomes. Inadequately treated disease may cause high morbidity, negatively impacting quality of life and leading to increased costs for supportive care. To address the unmet needs of these patients, we propose an exploratory trial combining Avelumab with radiation therapy, with an investigational plan to study clinical and health services outcomes. Cutaneous squamous cell carcinoma also represents a unique opportunity for correlative studies, given the accessibility of disease. The schedule of patient biopsies has been designed to allow analyses following treatment with Avelumab monotherapy as well as concurrent Avelumab/RT. We therefore propose additional biomarker outcomes, which may improve the care of patients with cuSCC as well as those with a host of solid tumors already sensitive to immunotherapy.

* Patients with cuSCC deemed unresectable (TxNxM0 - stage I-IV, M0);
* Prior to screening, patients will be reviewed at a bi-monthly multi-disciplinary cutaneous tumor board to determine unresectability; representatives from dermatology, pathology, medical oncology, radiation oncology, general surgery, and if deemed necessary, plastic surgery will be included;
* Patients must possess an Eastern Co-operative Oncology Group (ECOG) performance status ≤ 2 This study has been designed as an open-label, non-randomized, single-arm phase II study to investigate the feasibility and efficacy of Avelumab in combination with radiation therapy in patients with unresectable cuSCC.

All evaluable patients will be evaluated using identical instruments, and analysis will be by intent-to-treat. Toxicity will be assessed using standardized criteria (CTCAE version 4.03) by trained trial staff. Quality of life instruments will be administered to patients prior to their medical assessments. Every effort will be made to limit lost or missing data and incomplete follow-up.

Based on the primary objective of the study sample size of 20 patients is proposed.

This sample size calculation is based on the historical response rate associated with radiation therapy of 50%. The investigators predict an improvement in response using Avelumab and radiation therapy of 30%, in other words a net overall response rate of 80%. Utilizing a one-sided, binomial hypothesis test with a target p value of 0.05, the total sample size would be 18 to achieve a power of 80% for the study. The null hypothesis will be rejected if 13 out of 18 patients demonstrate an objective tumor response following treatment, indicating further study is warranted. Assuming a dropout rate of 10% (patient dropout defined as voluntary withdrawal from active therapy prior to completion of treatment), an additional 2 patients would have to be enrolled, bringing the total target enrollment to 20 patients.

The total duration of accrual is anticipated to last 26 months. With a maximum follow-up of 24 months following treatment of the eighteenth patient enrolled to study, the maximum study duration is not anticipated to exceed 50 months.

The provision of a tumor biopsy is optional, but strongly encouraged. For those patients who consent to tumor biopsy, samples (either punch, needle-core or shave-biopsy) will be obtained in advance of treatment, 2 weeks post first cycle of Avelumab (but before the initiation of radiation therapy) and in conjunction with the 30-day safety analysis.

An electronic data capture system will be used in this trial. A case report form (CRF) will have to be completed for each consented patient. The site maintains a separate source of data. This data will be entered by the site into the electronic data capture system This study is proposed as a phase II study with objective response rate as the primary endpoint. Refer to section 3.3.1 for the estimated calculation of study sample size.

If the study conduct (e.g. recruitment rate, drop-out rate, data quality, protocol compliance) does not suggest a proper completion of the study within a reasonable time frame the trial will be terminated. This will be done in consultation with the CCI DSMB.

The trial activities performed at the CCI will be monitored by the Cross Cancer Institute, Investigator Initiated Trials Data Safety Monitoring Board. The DSMB is independent of the investigator and is composed of representatives from both medical and radiation oncology. Further details about its charter can be found by contacting the Project Manager, Investigator Initiated Clinical Trials at the Cross Cancer institute.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 years of age or older.
2. Patients with histologically confirmed, unresectable cuSCC, stage I-IV (M0).
3. Patients must be capable of providing consent to enrolment and treatment.
4. Patients with a performance status of ECOG 0-2 will be eligible for enrolment
5. Measurable disease must be present according to RECIST 1.1 criteria.
6. Women of child bearing potential (WOCBP) must have a negative serum (or urine) pregnancy test at the time of screening. WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy or bilateral salpingectomy) and is not postmenopausal. Menopause is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes. In addition, females under the age of 55 years must have a serum follicle stimulating hormone, (FSH) level > 40 mIU/mL to confirm menopause.
7. Patients of childbearing / reproductive potential should use highly effective birth control methods, as defined by the investigator, during the study treatment period and for a period of 30 days after the last dose of study drug. A highly effective method of birth control is defined as those that result in low failure rate (i.e. less than 1% per year) when used consistently and correctly.

   Note: abstinence is acceptable if this is established and preferred contraception for the patient and is accepted as a local standard.
8. Female patients who are breast-feeding should discontinue nursing prior to the first dose of study treatment and until 30 days after the last dose of study drug.
9. Male patients should agree to not donate sperm during the study and for a period of at least 30 days after last dose of study drug.
10. Absence of any condition hampering compliance with the study protocol and follow- up schedule; those conditions should be discussed with the patient before registration in the trial.
11. The following adequate organ function laboratory values must be met:

Hematological:

* Absolute neutrophil count (ANC) >1.5 x109/L
* Platelet count >100 x109/L
* Hemoglobin >9 g/dL (may have been transfused)

Renal:

o Estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method)

Hepatic:

* Total serum bilirubin <1.5x ULN
* AST and ALT <2.5x ULN

Coagulation:

* International Normalized Ratio (INR) <1.5x ULN (unless patient is receiving anticoagulant therapy as long as prothrombin time (PT) or activated partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants)
* PTT <1.5x ULN (unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants)

Exclusion Criteria:

1. History of pneumonitis requiring treatment with steroids.
2. History of active interstitial lung disease.
3. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
4. History of another malignancy or a concurrent malignancy; Exceptions include patients who have been disease-free for 3 years, or patients with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible, for example cervical cancer in situ.
5. Diagnosis of immunodeficiency.
6. Current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
7. Prior organ transplantation including allogeneic stem-cell transplantation.
8. Known history of human immunodeficiency virus (HIV).
9. Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV ribonucleic acid (RNA) if anti-HCV antibody screening test positive).
10. Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
11. Active infection requiring systemic therapy.
12. Vaccination within 4 weeks of the first dose of Avelumab and while on trials is prohibited except for administration of inactivated vaccines.
13. Patient will not be eligible if the patient is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling or child) who is investigational site or sponsor staff directly involved with this trial, unless prospective independent ethics committee (IEC) approval (by chair or designee) is given allowing exception to this criterion for a specific subject.
14. Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (CTCAE v4.03 Grade ≥ 3).
15. Other severe acute or chronic medical conditions including inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
16. Persisting toxicity related to prior therapy (NCI CTCAE v. 4.03 grade > 1); however, alopecia, sensory neuropathy ≤ grade 2, or other toxicities ≤ grade 2 not constituting a safety risk based on investigator's judgment are acceptable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Objective response rate (assessing change in tumour response before treatment vs after) | Primary analysis to occur approximately 36 weeks after LPFV. Baseline staging at screening,repeated at 90 day fup and confirmatory scan
  Associated with combination Avelumab/radiation therapy (defined as the proportion of patients achieving either a partial response or a complete response as best-overall response per RECIST criteria 1.1)

SECONDARY OUTCOMES:
Progression-free survival | PFS will be based on the disease assessment or date of death provided by the investigator. The analysis of PFS will be scheduled to occur approximately 90 days following completion of the 24 month follow-up period for the final patient enrolled to study
  PFS is defined as the time between the date of treatment initiation and the date of disease progression (determined utilizing RECIST 1.1 criteria) or death (whatever the cause), whichever occurs first. For patients who remain alive and whose disease has not progressed, PFS data will be censored on the date of the last tumour assessment on study for patients who do not have objective tumour progression and who do not die while on study
Clinical and pathological response rate | The analysis of clinical and pathological response will be conducted within 90 days of enrollment of the last patient to study
  associated with Avelumab monotherapy (clinical response rate per RECIST 1.1; pathological response rate defined as the proportion of patients who, upon post-Avelumab monotherapy re-biopsy, demonstrate ≥ 10% increase tumor necrosis versus pre-treatment biopsy)
Safety analysis: CTCAE v.4.03 | Delegated study personnel will assess the patients for adverse events at baseline through to study completion per protocol (Baseline, cycles 1-5 (each cycle is 14 days), and in follow up at 30 days, 90 days and every 12 weeks up to 2 years).
  (treatment-related and non-related adverse events per CTCAE v.4.03)

OTHER OUTCOMES:
Utility of tumoral PD-L1 expression as a predictive and prognostic biomarker | Tumor biopsies will be obtained prior to treatment (baseline), following Avelumab monotherapy (post-cycle 1 treatment) and following completion of Avelumab concurrent with radiation therapy (end of cycle 4). Each cycle is 14 days.
  Quantitative immunohistochemical analysis of PD-L1 expression will be performed and correlated with treatment response. PD-L1 expression may be constitutive or inducible; radiation therapy has been demonstrated to induce the expression of PD-L1 on tumor cells(22). Tumor biopsy will be repeated during concurrent Avelumab/radiation treatment, and tumoral expression of PD-L1 analyzed.
Quantification/characterization of tumor-infiltrating lymphocytes/PBMCs | Blood samples will be obtained prior to treatment (baseline), after Avelumab monotherapy (post-cycle 1 treatment) following completion of Avelumab concurrent with radiation therapy (end of cycle 4). Each cycle is 14 days.
  To isolate TILs and collect PBMCs from this patient cohort according to the schedule in section 3.5.2 table 1.
Characterization of tumoral MHC-I/II expression/ Analysis of MHC immunopeptidomes | Tumor biopsies will be obtained prior to treatment (baseline), following Avelumab monotherapy (post-cycle 1 treatment) and following completion of Avelumab concurrent with radiation therapy. Each cycle is 14 days.
  The design of this study is such that pre- and post/during treatment biopsies can be compared for MHC antigen expression, hypothesizing that expression levels may have predictive value in the setting of checkpoint inhibition. Expression of MHC molecules (class I and class II) will be analyzed on pre- and post/during treatment biopsies by immunohistochemistry. In addition to quantifying tumoral expression of MHC I/II molecules at baseline, following treatment with Avelumab, and following treatment with Avelumab/RT, investigators propose small scale MHC class I immuno-isolation and peptide extraction(30) to determine the repertoire of antigenic peptides expressed at each of the three time-points. The investigators hypothesize that antigen quantity and diversity may have predictive value for response to Avelumab, and that treatment at each of the three time-points will alter the presentation of immunogenic antigens.
Patient-reported quality of life: Brief Older People's Quality of Life questionnaire (OPQOL-brief) | Assess patient-reported QoL at baseline and 30 days after last avelumab administration (cycle 5)
  Brief Older People's Quality of Life questionnaire (OPQOL-brief) will be used to assess patient-reported QoL.
  The OPQOL-BRIEF questionnaire has 13 items, with a preliminary single item on global QoL, shown below. This single item is not scored with the OPQOL; it is coded as Very good (1) to Very bad (5).
  Each of the 13 items is scored Strongly agree=1, Agree=2, Neither=3, Disagree=4, Strongly disagree=5. The items are summed for a total OPQOL-Brief score, then positive items are reverse coded, so that higher scores represented higher QoL.

CONTACTS AND LOCATIONS:
Overall Officials: John Walker, Walker, Principal Investigator — Alberta Health Services - Cross Cancer Institute
Locations (2):
- Canada (2):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta